CLINICAL TRIAL: NCT06380751
Title: A Randomised, Open-Label, Phase III Study of Saruparib (AZD5305) Plus Camizestrant Compared With Physician's Choice CDK4/6 Inhibitor Plus Endocrine Therapy or Plus Camizestrant for the First-Line Treatment of Patients With BRCA1, BRCA2, or PALB2 Mutations and Hormone Receptor Positive, HER2-Negative (IHC 0, 1+, 2+/ ISH Non-amplified) Advanced Breast Cancer (EvoPAR-Breast01)
Brief Title: Saruparib (AZD5305) Plus Camizestrant Compared With CDK4/6 Inhibitor Plus Endocrine Therapy or Plus Camizestrant in HR-Positive, HER2-Negative (IHC 0, 1+, 2+/ ISH Non-amplified), BRCA1, BRCA2, or PALB2m Advanced Breast Cancer
Acronym: EvoPAR-BR01
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D9722C00001
Record Dates: First submitted 2024-03-25; First posted 2024-04-24 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Advanced Breast Cancer
MeSH Terms: interventions — AZD5305; AZD9833; abemaciclib; ribociclib; palbociclib; Fulvestrant; Letrozole; Anastrozole; exemestane

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1: saruparib (AZD5305) plus camizestrant (Experimental): participants will receive saruparib (AZD5305) orally and camizestrant orally
  Interventions: Drug: Saruparib (AZD5305); Drug: Camizestrant
- Arm 2: Physician's choice CDK4/6i plus physician's choice ET (Active Comparator): agents are indicated below and should follow local guidelines:
  * Physician's Choice CDK4/6i:
    * abemaciclib orally, or
    * ribociclib orally, or
    * palbociclib orally.
  * Physician's Choice ET:
    * fulvestrant intramuscularly, or
    * One of the following AIs:
      * letrozole orally, or
      * anastrozole orally, or
      * exemestane orally
  Interventions: Drug: Abemaciclib; Drug: Ribociclib; Drug: Palbociclib; Drug: Fulvestrant; Drug: Letrozole; Drug: Anastrozole; Drug: Exemestane
- Arm 3: Physician's choice CDK4/6i plus camizestrant (Experimental): participants will receive camizestrant orally. Agents for CDK4/6i treatment are indicated above and should follow local guidelines
  Interventions: Drug: Camizestrant; Drug: Abemaciclib; Drug: Ribociclib; Drug: Palbociclib

INTERVENTIONS:
Drug: Saruparib (AZD5305) — Saruparib (AZD5305) is a potent and selective inhibitor of PARP1, with minimal effect on PARP2.
  Arms: Arm 1: saruparib (AZD5305) plus camizestrant
Drug: Camizestrant — Camizestrant (AZD9833) is an orally bioavailable, next generation SERD with non-clinical and clinical activity in both ESR1 mutant and wild type settings .
  Arms: Arm 1: saruparib (AZD5305) plus camizestrant; Arm 3: Physician's choice CDK4/6i plus camizestrant
Drug: Abemaciclib — CDK4/6 Inhibitor
  Arms: Arm 2: Physician's choice CDK4/6i plus physician's choice ET; Arm 3: Physician's choice CDK4/6i plus camizestrant
Drug: Ribociclib — CDK4/6 Inhibitor
  Arms: Arm 2: Physician's choice CDK4/6i plus physician's choice ET; Arm 3: Physician's choice CDK4/6i plus camizestrant
Drug: Palbociclib — CDK 4/6 Inhibitor
  Arms: Arm 2: Physician's choice CDK4/6i plus physician's choice ET; Arm 3: Physician's choice CDK4/6i plus camizestrant
Drug: Fulvestrant — Endocrine Therapy
  Arms: Arm 2: Physician's choice CDK4/6i plus physician's choice ET
Drug: Letrozole — Endorcine Therapy
  Arms: Arm 2: Physician's choice CDK4/6i plus physician's choice ET
Drug: Anastrozole — Endocrine Therapy
  Arms: Arm 2: Physician's choice CDK4/6i plus physician's choice ET
Drug: Exemestane — Endocrine Therapy
  Arms: Arm 2: Physician's choice CDK4/6i plus physician's choice ET

SUMMARY:
The primary objective of the study is to measure efficacy of saruparib (AZD5305) plus camizestrant compared with physician's choice CDK4/6i plus ET in patients with BRCA1, BRCA2, or PALB2m, HR-positive, HER2-negative (defined as IHC 0, 1+, 2+/ ISH non-amplified) advanced breast cancer

DETAILED DESCRIPTION:
Approximately 2,620 participants will be screened to achieve approximately 500 participants randomised to study intervention.

Participants will be randomised in a 2:2:1 ratio to one of the following intervention groups:

* Arm 1: saruparib (AZD5305) plus camizestrant
* Arm 2: Physician's choice CDK4/6i plus physician's choice ET
* Arm 3: Physician's choice CDK4/6i plus camizestrant Treatment continues until BICR-confirmed disease progression, unacceptable toxicity occurs, or the participant withdraws consent.

ELIGIBILITY:
Inclusion Criteria:

* Adult females, pre/peri-menopausal and/or post-menopausal, and adult males
* Histologically or cytologically documented diagnosis of HR-positive, HER2-negative breast cancer
* Advanced breast cancer with either locally advanced disease not amenable to curative treatment or metastatic disease
* ECOG performance status of 0 or 1 with no deterioration over the previous 2 weeks
* FFPE tumour tissue from each participant
* Documented germline tumour loss of function mutation in BRCA1, BRCA2, or PALB2
* Adequate organ and marrow function

Exclusion Criteria:

* Participants with history of MDS/AML or with features suggestive of MDS/AML
* Participants with any known predisposition to bleeding
* Any history of persisting severe cytopenia
* Any evidence of severe or uncontrolled systemic diseases or active uncontrolled infections
* Refractory nausea and vomiting, chronic GI disease, inability to swallow the formulated product, or previous significant bowel resection
* History of another primary malignancy
* Persistent toxicities (CTCAE Grade ≥ 2) caused by previous anti-cancer therapy excluding alopecia
* Spinal cord compression, brain metastases, carcinomatous meningitis, or leptomeningeal disease
* Evidence of active and uncontrolled hepatitis B and/or hepatitis C
* Evidence of active and uncontrolled HIV infection
* Active tuberculosis infection
* Cardiac criteria, including history of arrythmia and cardiovascular disease
* Concurrent exogenous reproductive hormone therapy or non-topical hormonal therapy for non-cancer-related conditions
* Major surgical procedure or significant traumatic injury within 4 weeks of the first dose of study intervention or an anticipated need for major surgery during the study
* Palliative radiotherapy with a limited field of radiation within 2 weeks or with wide field of radiation or to more than 30% of the bone marrow within 4 weeks before the first dose of study treatment
* Prior treatment with systemic anti-cancer therapy for locoregionally recurrent or metastatic disease is not permitted, apart from treatment with ET up to 28 days before randomisation
* Prior treatment within 28 days with blood product support or growth factor support
* Any systemic concurrent anti-cancer treatment
* Concomitant use of the following types of medications or herbal supplements within 21 days or at least 5 half-lives of randomisation:

  1. Strong and moderate CYP3A4 inducers/inhibitors
  2. Sensitive CYP2B6 substrates
  3. Substrates of CYP2C9 and/or CYP2C19 which have a narrow therapeutic index, eg, warfarin (and other coumarin-derived vitamin K antagonist anticoagulants) and phenytoin.
* Concomitant use of drugs that are known to prolong QT and have a known risk of TdP
* Systemic use of atropine
* The following exclusion criteria apply to treatments administered for early breast cancer:

  1. Disease progression ≤ 84 days following the last dose of neo-adjuvant or adjuvant chemotherapy
  2. Disease progression ≤ 1 year (365 days) from the last dose of treatment with a PARPi and/or platinum agent for early breast cancer
  3. Disease progression ≤ 1 year (365 days) from the last dose with a CDK4/6i in the adjuvant setting
  4. Disease progression ≤ 1 year (365 days) from the last dose of an oral SERD including camizestrant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2029-03-30 (Estimated); Study Completion 2030-10-18 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | Up to approximately 59 months
  PFS is defined as time from randomisation until progression per RECIST v1.1 as assessed by BICR, or death due to any cause.

SECONDARY OUTCOMES:
Overall Survival | Up to approximately 88 months
  OS is defined as the time from randomisation until the date of death due to any cause.
Progression Free Survival 2 | Up to approximately 59 months
  PFS2 is defined as the time from randomisation to the earliest of the progression event (following the initial investigator-assessed progression), after first subsequent therapy, or death.
Time to chemotherapy | Up to approximately 59 months
  Time to chemotherapy is defined as time from randomisation until the start date of the first subsequent chemotherapy treatment after discontinuation of randomised treatment (censoring participants who died prior to initiation of chemotherapy).
Objective Response Rate | Up to approximately 59 months
  ORR is defined as the proportion of participants who have a complete or parial response, as determined by BICR per RECIST v1.1.
Duration of Response | Up to approximately 59 months
  DoR is defined as the time from the date of first documented response until date of documented progression per RECIST v1.1 as assessed by BICR, or death due to any cause.
Participant-reported tolerability | Up to approximately 59 months
  Proportion of all dosed participants reporting different levels of severity of diarrhoea as measured by the diarrhoea single item (EORTC IL237/IL239/IL240) and different levels of severity of abdominal pain as measured by the abdominal pain single item (EORTC IL237/IL239/IL240).
Time to deterioration in patient-reported global health status/QoL as measured by the global health status/QoL scale within the The European Organisation for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ) | Up to approximately 59 months
  This scale includes 2 items asking participants to report overall health and overall quality of life in the past week. Both items are measured on a 6-point verbal rating scale ranging from Very Poor to Excellent. Single item scores are averaged to calculate a subscale score that is transformed to range from 0 to 100, where higher scores indicate better global health status/QoL.
Change from baseline in patient-reported global health status/QoL as measured by the global health status/QoL scale within the The European Organisation for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ) | Up to approximately 59 months
  This scale includes 2 items asking participants to report overall health and overall quality of life in the past week. Both items are measured on a 6-point verbal rating scale ranging from Very Poor to Excellent. Single item scores are averaged to calculate a subscale score that is transformed to range from 0 to 100, where higher scores indicate better global health status/QoL.
Plasma concentrations of saruparib (AZD5305) | Up to approximately 59 months
Plasma concentrations of camizestrant | Up to approximately 59 months
Samples will be used to develop companion diagnostics by analyzing their performance characteristics and calculate their consistency with clinical trial assays used for enrolment onto the study. | Up to approximately 59 months
  Samples will be tested by a CDx to confirm BRCA1/2 and PALB2 gene mutation status

CONTACTS AND LOCATIONS:
Locations (245):
- United States (45):
  - Research Site, Gilbert, Arizona
  - Research Site, Fountain Valley, California
  - Research Site, Glendale, California
  - Research Site, Los Angeles, California
  - Research Site, Newport Beach, California
  - Research Site, Aurora, Colorado
  - Research Site, Grand Junction, Colorado
  - Research Site, Hollywood, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Orlando, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Evanston, Illinois
  - Research Site, Park Ridge, Illinois
  - Research Site, Urbana, Illinois
  - Research Site, Winfield, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Louisville, Kentucky
  - Research Site, Silver Spring, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Dearborn, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, Royal Oak, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, Springfield, Missouri
  - Research Site, Camden, New Jersey
  - Research Site, New Brunswick, New Jersey
  - Research Site, Brooklyn, New York
  - Research Site, Mineola, New York
  - Research Site, New Hyde Park, New York
  - Research Site, New York, New York
  - Research Site, Shirley, New York
  - Research Site, Stony Brook, New York
  - Research Site, The Bronx, New York
  - Research Site, Westbury, New York
  - Research Site, Hershey, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, West Columbia, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Norfolk, Virginia
  - Research Site, Tacoma, Washington
  - Research Site, Morgantown, West Virginia
  - Research Site, Milwaukee, Wisconsin
- Argentina (6):
  - Research Site, Ciudad Autónoma Buenos Aires
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Córdoba
  - Research Site, Rosario
  - Research Site, Salta
  - Research Site, San Miguel de Tucumán
- Australia (3):
  - Research Site, Darlinghurst
  - Research Site, Malvern
  - Research Site, Melbourne
- Austria (4):
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Linz
  - Research Site, Vienna
- Brazil (9):
  - Research Site, Cachoeira de Itapemirim
  - Research Site, Curitiba
  - Research Site, Fortaleza
  - Research Site, Goiânia
  - Research Site, Jaú
  - Research Site, Porto Alegre
  - Research Site, Ribeirão Preto
  - Research Site, Salvador
  - Research Site, São Paulo
- Bulgaria (4):
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Stara Zagora
  - Research Site, Vratsa
- Canada (5):
  - Research Site, Toronto, Ontario
  - Research Site, Greenfield Park, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Saskatoon, Saskatchewan
  - Research Site, Toronto
- Chile (5):
  - Research Site, Providencia
  - Research Site, Recoleta
  - Research Site, Santiago
  - Research Site, Talca
  - Research Site, Viña del Mar
- China (31):
  - Research Site, Beijing
  - Research Site, Bengbu
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Foshan
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Hohhot
  - Research Site, Jining
  - Research Site, Kunming
  - Research Site, Liuchow
  - Research Site, Luoyang
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Shandong
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shijiazhuang
  - Research Site, Tianjin
  - Research Site, Weifang
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Xiamen
  - Research Site, Xiangfan
  - Research Site, Xinxiang
  - Research Site, Zhengzhou
- Czechia (5):
  - Research Site, Brno
  - Research Site, Hořovice
  - Research Site, Hradec Králové
  - Research Site, Olomouc
  - Research Site, Prague
- France (10):
  - Research Site, Angers
  - Research Site, Besançon
  - Research Site, Lille
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Paris
  - Research Site, Rouen
  - Research Site, Saint-Herblain
  - Research Site, Toulouse
  - Research Site, Villejuif
- Germany (16):
  - Research Site, Aachen
  - Research Site, Augsburg
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Dessau
  - Research Site, Düsseldorf
  - Research Site, Erlangen
  - Research Site, Göttingen
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Kiel
  - Research Site, Leipzig
  - Research Site, Ludwigsburg
  - Research Site, München
  - Research Site, Münster
- Research Site, Hong Kong, Hong Kong
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Miskolc
  - Research Site, Zalaegerszeg
- India (10):
  - Research Site, Delhi
  - Research Site, Kolkata
  - Research Site, Lucknow
  - Research Site, Mumbai
  - Research Site, Mysuru
  - Research Site, Nagpur
  - Research Site, Nashik
  - Research Site, New Delhi
  - Research Site, Surat
  - Research Site, Thiruvananthapuram
- Israel (4):
  - Research Site, Jerusalem
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
  - Research Site, Tel Aviv
- Italy (9):
  - Research Site, Bergamo
  - Research Site, Bologna
  - Research Site, Milan
  - Research Site, Modena
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Reggio Emilia
  - Research Site, Rome
  - Research Site, Rozzano
- Japan (21):
  - Research Site, Chiba
  - Research Site, Hidaka-shi
  - Research Site, Hirakata-shi
  - Research Site, Isehara-shi
  - Research Site, Kagoshima
  - Research Site, Kashiwa
  - Research Site, Kōtoku
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Matsuyama
  - Research Site, Nagoya
  - Research Site, Osaka
  - Research Site, Ota-shi
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Shinagawa-ku
  - Research Site, Suita-shi
  - Research Site, Sunto-gun
  - Research Site, Takasaki-shi
  - Research Site, Tsu
  - Research Site, Yokohama
- Malaysia (5):
  - Research Site, Bandar Puncak Alam
  - Research Site, Johor Bahru
  - Research Site, Kuala Lumpur
  - Research Site, Kuala Selangor
  - Research Site, Malacca
- Peru (3):
  - Research Site, Bellavista
  - Research Site, Jesus Maria, Lima
  - Research Site, Lima
- Poland (5):
  - Research Site, Biała Podlaska
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Poznan
  - Research Site, Warsaw
- Portugal (5):
  - Research Site, Coimbra
  - Research Site, Lisbon
  - Research Site, Matosinhos Municipality
  - Research Site, Porto
  - Research Site, Vila Real
- Research Site, San Juan, Puerto Rico
- South Korea (3):
  - Research Site, Daegu
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (9):
  - Research Site, Barcelona
  - Research Site, Cáceres
  - Research Site, Granada
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Pamplona
  - Research Site, Seville
  - Research Site, Valencia
- Taiwan (5):
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (4):
  - Research Site, Bangkok
  - Research Site, Dusit
  - Research Site, Hat Yai
  - Research Site, Ratchathewi
- Turkey (Türkiye) (5):
  - Research Site, Adapazarı
  - Research Site, Altındağ-Ankara
  - Research Site, Çankaya
  - Research Site, Istanbul
  - Research Site, Kayseri
- United Kingdom (8):
  - Research Site, Cambridge
  - Research Site, Guildford
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Oxford
  - Research Site, Swansea
  - Research Site, Taunton
  - Research Site, Truro

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home